CLINICAL TRIAL: NCT06500754
Title: Study of the Causes and Consequences of Persistent Villous Atrophy Despite an Intentionally Strict Gluten-free Diet in Celiac Disease Patients - Effect of an Ultra-strict Gluten-free Diet on Persistent Villous Atrophy
Brief Title: Persistent Villous Atrophy in Celiac Disease Patients Following an Intentionally Strict Gluten-free Diet
Acronym: CADER2
Status: Recruiting | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: P/21-098
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Celiac Disease; Villous Atrophy of Intestine
Keywords: persistent villous atrophy; ultra-strict gluten-free diet; microbiota; epigenetics
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — duodenal biopsy samples, blood, urine and feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Celiac Disease patients
  Interventions: Other: Ultra-strict gluten-free diet

INTERVENTIONS:
Other: Ultra-strict gluten-free diet — ultra-strict gluten-free diet (avoiding traces and contamination) under dietitian supervision

SUMMARY:
Celiac disease (CD) is an immune-mediated disease characterized by small intestinal inflammation from gluten ingestion, a group of proteins present in various cereals, including wheat, rye, barley, spelt, and kamut. CD is the most common chronic gastrointestinal disease and one of the most common autoimmune disorders, estimated to affect 0.4-1.7% of the general population. Currently, a strict lifelong gluten-free diet (GFD) is the only available treatment to avoid the inappropriate inflammatory response and prevent the shortening of the villi lining the small intestine (villous atrophy). However, a significant proportion of CD patients, ranging from 4% to 79%, show persistent villous atrophy despite following an intentional GFD. The causative factors and the clinical consequences of persistent villous atrophy in CD patients are not well known yet but might resemble untreated CD long-term complications.

Interestingly, in the precedent study (CADER) persistent villous atrophy was found to be more present in patients diagnosed at an older age (65% of CD patients diagnosed after 30 years of age) than in younger patients. Moreover, unintentional exposure to gluten was found in 70% of the cases. The causative factors of this hypersensitivity to small amounts of gluten present in older patients are unknown. The intestinal microbiota and age-related epigenetic changes may help maintaining the dysregulation of the immune response, causing older patients to be hypersensitive to small amounts of gluten.

The aim of this study (CADER2) is to identify the immunological and clinical consequences of persistent villous atrophy in CD and study whether changes in the intestinal microbiome and age-related epigenetic modifications may contribute to it. Last, the investigators want to assess if an ultra-strict GFD can be a viable and effective alternative to treat this subset of CD patients. In order to achieve these objectives, the study includes 2 phases: 1) Cross-sectional study to assess the causes and the clinical consequences of persistent villous atrophy in CD patients; and 2) Longitudinal study to evaluate the potential therapeutic effect of an ultra-strict GFD on persistent villous atrophy and its subtle clinical manifestations.

The investigators hypothesize that persistent villous atrophy in CD patients despite an intentional GFD is associated with chronic low-grade inflammation and increased circulating cytokines in blood, potentially leading to cognitive deficits, fatigue, anxiety, depression, malnutrition, sarcopenia and osteoporosis. The intestinal microbiota and age-related epigenetic changes may help to maintain the dysregulation of the immune response, causing patients to be hypersensitive to small amounts of gluten. This subset of CD patient could highly benefit from an ultra-strict GFD.

To date, six centers have been recruited: Hospital Universitari Mutua Terrassa (Barcelona), Hospital Clínico San Carlos (Madrid), Hospital Fundación Jiménez Díaz (Madrid), Hospital Universitario de La Princesa (Madrid), Hospital Universitario Ramón y Cajal (Madrid) and Hospital Universitario Virgen Macarena (Sevilla). Digestive, endocrine, nutritional and clinical psychology experts will be involved in the monitoring of the patients. Microbiome analysis will be performed at the Genomics Unit, Microbiota Laboratory (LABMIC) of the IdISSC (Madrid). The methylation studies (age-related epigenetic modifications) will be hired externally.

Overall, the results of this study (CADER2) may help identify new therapeutic strategies as well as improve the management of chronicity and care of CD patients who do not respond to the current treatment. Furthermore, it will contribute to a deeper understanding of the pathophysiological relationships between diet, microbiome, genetics and immunology in CD.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis 18 years or more.
* Diagnosis of CD with villous atrophy, positive serology and clinical and serological response to GFD.
* To be in a GFD for at least 2 years, with good adherence to it.
* Negative or positive anti-transglutaminase (tTG2) IgA antibodies at low titers (<2 times the normal value) at recruitment.
* Written informed consent.

Exclusion Criteria:

* Refractory CD (RCD) type 2 and type 1
* Other associated intestinal diseases (inflammatory bowel disease, microscopic colitis, other types of enteropathies).
* Need for treatment with corticosteroids or immunosuppressants.
* Surgeries or other diseases predisposing to bacterial overgrowth in the small intestine.
* Pregnancy, lactation.
* Associated chronic diseases (lung, heart, kidney, liver cirrhosis).
* Alcoholism or drug addiction.
* Schizophrenia-type psychiatric diseases, other psychoses, bipolar.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Celiac Disease patients from the participating hospitals
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Persistent villous atrophy frequency | at inclusion
  proportion of patients showing villous atrophy after 2 years of an intentionally strict gluten-free diet

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari MútuaTerrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Fernandez-Banares F, Beltran B, Salas A, Comino I, Ballester-Clau R, Ferrer C, Molina-Infante J, Rosinach M, Modolell I, Rodriguez-Moranta F, Arau B, Segura V, Fernandez-Salazar L, Santolaria S, Esteve M, Sousa C; CADER study group. Persistent Villous Atrophy in De Novo Adult Patients With Celiac Disease and Strict Control of Gluten-Free Diet Adherence: A Multicenter Prospective Study (CADER Study). Am J Gastroenterol. 2021 May 1;116(5):1036-1043. doi: 10.14309/ajg.0000000000001139. PMID 33491958
- [Background] Catassi C, Fabiani E, Iacono G, D'Agate C, Francavilla R, Biagi F, Volta U, Accomando S, Picarelli A, De Vitis I, Pianelli G, Gesuita R, Carle F, Mandolesi A, Bearzi I, Fasano A. A prospective, double-blind, placebo-controlled trial to establish a safe gluten threshold for patients with celiac disease. Am J Clin Nutr. 2007 Jan;85(1):160-6. doi: 10.1093/ajcn/85.1.160. PMID 17209192
- [Background] Collin P, Maki M, Kaukinen K. Safe gluten threshold for patients with celiac disease: some patients are more tolerant than others. Am J Clin Nutr. 2007 Jul;86(1):260; author reply 260-1. doi: 10.1093/ajcn/86.1.260. No abstract available. PMID 17616789
- [Background] Hollon JR, Cureton PA, Martin ML, Puppa EL, Fasano A. Trace gluten contamination may play a role in mucosal and clinical recovery in a subgroup of diet-adherent non-responsive celiac disease patients. BMC Gastroenterol. 2013 Feb 28;13:40. doi: 10.1186/1471-230X-13-40. PMID 23448408
- [Background] Sharkey LM, Corbett G, Currie E, Lee J, Sweeney N, Woodward JM. Optimising delivery of care in coeliac disease - comparison of the benefits of repeat biopsy and serological follow-up. Aliment Pharmacol Ther. 2013 Nov;38(10):1278-91. doi: 10.1111/apt.12510. Epub 2013 Oct 5. PMID 24117503
- [Background] Lebwohl B, Michaelsson K, Green PH, Ludvigsson JF. Persistent mucosal damage and risk of fracture in celiac disease. J Clin Endocrinol Metab. 2014 Feb;99(2):609-16. doi: 10.1210/jc.2013-3164. Epub 2014 Jan 16. PMID 24432993
- [Background] Lebwohl B, Granath F, Ekbom A, Smedby KE, Murray JA, Neugut AI, Green PH, Ludvigsson JF. Mucosal healing and risk for lymphoproliferative malignancy in celiac disease: a population-based cohort study. Ann Intern Med. 2013 Aug 6;159(3):169-75. doi: 10.7326/0003-4819-159-3-201308060-00006. PMID 23922062
- [Background] Kaukinen K, Peraaho M, Lindfors K, Partanen J, Woolley N, Pikkarainen P, Karvonen AL, Laasanen T, Sievanen H, Maki M, Collin P. Persistent small bowel mucosal villous atrophy without symptoms in coeliac disease. Aliment Pharmacol Ther. 2007 May 15;25(10):1237-45. doi: 10.1111/j.1365-2036.2007.03311.x. PMID 17451570
- [Background] Manavalan JS, Hernandez L, Shah JG, Konikkara J, Naiyer AJ, Lee AR, Ciaccio E, Minaya MT, Green PH, Bhagat G. Serum cytokine elevations in celiac disease: association with disease presentation. Hum Immunol. 2010 Jan;71(1):50-7. doi: 10.1016/j.humimm.2009.09.351. PMID 19735687
- [Background] Heydari F, Rostami-Nejad M, Moheb-Alian A, Mollahoseini MH, Rostami K, Pourhoseingholi MA, Aghamohammadi E, Zali MR. Serum cytokines profile in treated celiac disease compared with non-celiac gluten sensitivity and control: a marker for differentiation. J Gastrointestin Liver Dis. 2018 Sep;27(3):241-247. doi: 10.15403/jgld.2014.1121.273.hey. PMID 30240467
- [Background] Dunne MR, Byrne G, Chirdo FG, Feighery C. Coeliac Disease Pathogenesis: The Uncertainties of a Well-Known Immune Mediated Disorder. Front Immunol. 2020 Jul 8;11:1374. doi: 10.3389/fimmu.2020.01374. eCollection 2020. PMID 32733456
- [Background] Olano C, Lopez V, Freire T, Rodriguez X, Pontet Y, Aleman A, Rodriguez N, Rovira L, Trucco E, Osinaga E, Cohen H, Quigley EM. Irritable bowel syndrome in celiac disease - relationships to celiac disease antibodies and levels of pro-inflammatory cytokines. Rev Gastroenterol Peru. 2020 Apr-Jun;40(2):127-135. PMID 32876628
- [Background] Yelland GW. Gluten-induced cognitive impairment ("brain fog") in coeliac disease. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:90-93. doi: 10.1111/jgh.13706. PMID 28244662
- [Background] Makhlouf S, Messelmani M, Zaouali J, Mrissa R. Cognitive impairment in celiac disease and non-celiac gluten sensitivity: review of literature on the main cognitive impairments, the imaging and the effect of gluten free diet. Acta Neurol Belg. 2018 Mar;118(1):21-27. doi: 10.1007/s13760-017-0870-z. Epub 2017 Dec 15. PMID 29247390
- [Background] Croall ID, Tooth C, Venneri A, Poyser C, Sanders DS, Hoggard N, Hadjivassiliou M. Cognitive Impairment in Coeliac Disease with Respect to Disease Duration and Gluten-Free Diet Adherence: A Pilot Study. Nutrients. 2020 Jul 8;12(7):2028. doi: 10.3390/nu12072028. PMID 32650524
- [Background] Croall ID, Sanders DS, Hadjivassiliou M, Hoggard N. Cognitive Deficit and White Matter Changes in Persons With Celiac Disease: A Population-Based Study. Gastroenterology. 2020 Jun;158(8):2112-2122. doi: 10.1053/j.gastro.2020.02.028. Epub 2020 Feb 20. PMID 32088203
- [Background] Tuttle CSL, Thang LAN, Maier AB. Markers of inflammation and their association with muscle strength and mass: A systematic review and meta-analysis. Ageing Res Rev. 2020 Dec;64:101185. doi: 10.1016/j.arr.2020.101185. Epub 2020 Sep 26. PMID 32992047
- [Background] Ciudin A, Simo-Servat A, Palmas F, Barahona MJ. Sarcopenic obesity: a new challenge in the clinical practice. Endocrinol Diabetes Nutr (Engl Ed). 2020 Dec;67(10):672-681. doi: 10.1016/j.endinu.2020.03.004. Epub 2020 Jun 18. English, Spanish. PMID 32565081
- [Background] Capriles VD, Martini LA, Areas JA. Metabolic osteopathy in celiac disease: importance of a gluten-free diet. Nutr Rev. 2009 Oct;67(10):599-606. doi: 10.1111/j.1753-4887.2009.00232.x. PMID 19785691
- [Background] Ray D, Yung R. Immune senescence, epigenetics and autoimmunity. Clin Immunol. 2018 Nov;196:59-63. doi: 10.1016/j.clim.2018.04.002. Epub 2018 Apr 11. PMID 29654845